CLINICAL TRIAL: NCT03125642
Title: Autologous Stem Cell Transplant In Patients With Hodgkin Lymphoma (HL) and Non-Hodgkin Lymphomas (NHL)
Brief Title: Auto Stem Cell Transplant for Lymphoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS132; MT2016-11C (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Lymphoblastic Lymphoma; Mature B-cell Lymphomas; Follicular Lymphoma; Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma; Burkitt's/Burkitt's like; Mature T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, T-Cell | interventions — Etoposide; Carmustine; Cytarabine; Melphalan; Peripheral Blood Stem Cell Transplantation; Granulocyte Colony-Stimulating Factor; Filgrastim; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- BEAM: NHL & HL (Experimental): BCNU, etoposide, Ara-C and melphalan (BEAM) for all NHL and those HL patients who are unable to receive CBV
  Interventions: Drug: Etoposide; Drug: BCNU; Drug: AraC; Drug: Melphalan; Procedure: Peripheral blood stem cell transplantation; Biological: G-CSF
- CBV: HL (Experimental): Cyclophosphamide, BCNU and VP-16 (CBV) for HL patients
  Interventions: Drug: Etoposide; Drug: BCNU; Drug: Cyclophosphamide
- CY/TBI (Experimental): Cyclophosphamide/Total Body Irradiation (CY/TBI) for patients with recent history of CNS lymphoma or those with allergies/contra-indications to agents used in BEAM
  Interventions: Procedure: Peripheral blood stem cell transplantation; Biological: G-CSF; Drug: Cyclophosphamide; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Etoposide — BEAM: 100 mg/m^2 IV over 2 hours BID on Days -5, -4, -3, -2 | CBV: 150 mg/m^2 intravenously over 4 hours every 12 hours starting at 6 a.m. and 6 p.m. on Days -6, -5, -4
  Other Names: VP-16
  Arms: BEAM: NHL & HL; CBV: HL
Drug: BCNU — BEAM & CBV: 300 mg/m^2 IV over over 2 hours on Day -6
  Other Names: Carmustine
  Arms: BEAM: NHL & HL; CBV: HL
Drug: AraC — BEAM: 100 mg/m^2 IV over 1 hour BID on Days -5, -4, -3, -2
  Other Names: Cytarabine; cytosine arabinoside; Cytosar-U; Depocyt
  Arms: BEAM: NHL & HL
Drug: Melphalan — BEAM: 140 mg/m^2 IV over 20 minutes on Day -1
  Other Names: Alkeran
  Arms: BEAM: NHL & HL
Procedure: Peripheral blood stem cell transplantation — All Arms: Day 0 infuse PBSC. All patients will have PBSC collected by leukapheresis. Mobilization will be done with G-CSF.
  Other Names: PBSC
  Arms: BEAM: NHL & HL; CY/TBI
Biological: G-CSF — All patients should receive G-CSF, 5 ug/kg/day IV as a bolus injection each evening beginning on day +5 until the ANC is >2500 x 10^9/L for 2 consecutive days. G-CSF will subsequently be restarted at 5 ug/kg/day SC or IV if the ANC falls below 1000/mm^3
  Other Names: filgrastim
  Arms: BEAM: NHL & HL; CY/TBI
Drug: Cyclophosphamide — CBV: 1.5 gm/M^2 over 2 hours at 10 a.m. on Days -6, -5, -4, -3 | CY/TBI: 60 mg/kg IV over 2 hours on Days -7, -6
  Other Names: Cytoxan
  Arms: CBV: HL; CY/TBI
Radiation: Total Body Irradiation — CY/TBI: 165 cGy bid on Day -4, -3, -2, -1
  Other Names: TBI
  Arms: CY/TBI

SUMMARY:
This is a phase II study of autologous transplant for patients with Hodgkin (HL) and non-Hodgkin lymphomas (NHL) including those who are HIV positive.

ELIGIBILITY:
Inclusion Criteria:

* Eligible Diseases

  1. Non-Hodgkin's Lymphoma (NHL)

     * Patients with chemo-sensitive histologically confirmed NHL will be eligible for this treatment protocol contingent on histologic sub-classification.
     * Patients in partial or complete remission following cell therapy will also be eligible.
     * NHL patients with resistant or refractory lymphoma (no PR following up to three cycles of combination chemotherapy) will not be eligible for transplant in this trial.
     * Lymphoblastic Lymphoma:

       1. All patients will be eligible in second or greater complete remission (CR) or first or subsequent partial remission (PR)
       2. Patients with any high-risk features will be eligible in first complete remission
       3. High risk features include: Stage IV, LDH >2 x upper limit of normal, ≥ 2 extranodal sites
     * Mature B-cell Lymphoma

       1. Follicular Lymphoma and other indolent lymphoma in ≥ second CR2/PR2
       2. Diffuse Large B-Cell Lymphoma: in ≥ CR2 or ≥ PR1; a high intermediate or high IPI (≥ 2 for age-adjusted IPI or ≥3 for IPI) at diagnosis and double-hit or triple-hit lymphoma will be eligible in first CR; transformed lymphoma from FL (or other indolent lymphoma) or chronic lymphocytic leukemia will be eligible if chemosensitive and bone marrow is negative
       3. Mantle Cell Lymphoma: in first or greater CR or PR
       4. Burkitt's/Burkitt's like: all patients except localized lymphoma will be eligible any time after initial therapy (after achievement of first complete remission), or in partial remission if they fail to achieve CR; patients with localized (stage I or Ziegler stage A) will be eligible only if they fail to achieve CR1 or after relapse
     * Mature T-Cell Lymphoma

       1. Chemosensitive T-cell lymphomas including Primary T-cell not otherwise specified angioimmunoblastic, and ALK-positive anaplastic large cell, will be eligible after initial therapy, whether or not CR is achieved.
       2. Mycosis fungoides/Sezary syndrome will be eligible in ≥CR2/PR2
  2. Hodgkin Lymphoma (HL)

     * Patients with histologically proven HL will be eligible for transplantation after failing prior therapy.
     * Patients with resistant disease (initial or at relapse): those who fail to achieve an objective partial response to three cycles of combination non-cross resistant chemotherapy will not be eligible for transplant in this trial.
     * For stage I/II patients treated with primary chemotherapy-radiation, they must have failed (no CR or progression after CR) at least one salvage combination chemotherapy treatment regimen
     * For advanced (stage III/IV) Hodgkin disease, patients must have failed an Adriamycin containing regimen (ABVD) or an alternative non-cross resistant regimen (e.g. MOPP)
     * Patients with any high-risk features will also be eligible, including those who:

       1. fail to achieve complete remission with initial combination chemotherapy
       2. have bulky disease after initial therapy (chemotherapy or radiation) defined as residual mediastinal mass ≥ 5 cm or other residual mass ≥ 10 cm accompanied by other features of persisting disease (e.g., PET scan positive; high LDH; enlarging on serial x-rays or biopsy positive) will be eligible - if feasible, persistent disease should be proven by biopsy
     * Patients should receive chemotherapy to attempt to achieve CR or minimal disease state for all patients pre-transplantation. The use of up to three cycles of non-cross resistant combination chemotherapy is advised.
     * Residual areas of limited disease should be considered for radiotherapy after and not prior to transplantation.
  3. HIV positive patients who are otherwise eligible for this study may be enrolled if they meet the following requirements:

     * Are seen in the infectious disease (ID)/HIV clinic prior to enrollment on study for the purpose of determining eligibility and for local coordination of HIV care during the peri-transplant period.
     * Are on maximally active anti-HIV regimen to control disease as determined appropriate by the ID/HIV physicians. For the majority of patients, this will be a highly active anti-retroviral therapy (HAART)-type therapy including a protease inhibitor.
     * CD4+ ≥ 50/µL
     * HIV RNA viral load ≤ 100,000 copies per mL on each of samples 4 weeks apart. The most recent level must be within 30 days of enrollment.
* Performance Status: Karnofsky Performance Status ≥ 80% for patients ≥ 16 years of age or Lansky Play Score ≥ 80 for patients < 16 years of age. Note: if poor performance status is due to lymphoma - KPS ≥ 60% or LPS ≥ 60 is acceptable
* Organ Function

  1. No evidence of serious organ dysfunction that is not attributable to tumor including:
  1. Hematologic:

     * hemoglobin > 8 gm/dL
     * WBC > 2.5 x 109/L with an ANC > 1.5 x 109/L off G-CSF or GM-CSF for 10 days or Neulasta for 21 days
     * platelets > 100 x 109/L without transfusion
     * bone marrow cellularity of > 20% with <5% involvement with tumor
  2. Renal: GFR > 50 ml/min/1.73m2 or serum creatinine ≤ 2.5 x ULN for age
  3. Hepatic: no history of severe prior or ongoing chronic liver disease. Total bilirubin ≤ 2.0 mg/dl, AST and alkaline phosphatase <5x upper limit of normal
  4. Cardiac: free of symptoms of uncontrolled cardiac disease including unstable angina, decompensated congestive heart failure, or arrhythmia. The ejection fraction by gated cardiac blood flow scan (MUGA) or Echocardiogram must be >40%
  5. Pulmonary: no significant obstructive airways disease (FEV1 must be ≥ 50%) and must have acceptable diffusion capacity (corrected DLCO > 50% of predicted)
  6. Central Nervous System: Patients with a history of CNS involvement by lymphoma or with relapsed primary CNS lymphoma will be eligible for Cy/TBI arm. Patients with active CNS disease are eligible if they have completed a standard treatment for CNS lymphoma and have no evidence of progressive CNS disease at the time of enrollment
* Other Inclusion Criteria

  1. At least 4 weeks from previous chemotherapy; 6 weeks from nitrosoureas
  2. Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment
  3. Patients who are carriers of Hepatitis B will be included in this study
  4. Voluntary written consent

Exclusion Criteria:

* Pregnant or breastfeeding: Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy
* Eligible for any higher priority transplant protocols
* Chemotherapy resistant disease
* Unrelated active infection

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Comparison | 3 years post transplant
  Compare progression-free survival (PFS) at 3 years post-transplant for patients who received who received a radiation free preparative regimen to the prior study MT2004-24 where NHL subjects received total body irradiation (TBI) as part of their preparative regimen.

SECONDARY OUTCOMES:
Overall Survival | 3 years post transplant
  Incidence of survival
Treatment related mortality | 6 months post transplant
  Incidence of treatment related mortality
Treatment related mortality | 1 year post transplant
  Incidence of treatment related mortality
Secondary malignancies | 3 years post transplant
  Cumulative incidence of secondary malignancies
Neutrophil engraftment | Day +1 to engraftment
  Average days to neutrophil engraftment
Platelet engraftment | Day +1 to engraftment
  Average days to platelet engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States